CLINICAL TRIAL: NCT00786981
Title: Epidural Steroid Injection Versus Epidural Steroid Injection and Manual Physical Therapy and Exercise in the Management of Lumbar Spinal Stenosis; a Randomized Clinical Trial
Brief Title: Epidural Steroid Injection Versus Epidural Steroid Injection and Manual Physical Therapy and Exercise in the Management of Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Joshua Cleland, DPT, OCS, Professor, Franklin Pierce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FP-36472
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural steroid injection and physical therapy (Other)
  Interventions: Other: Epidural steroid injection plus physical therapy
- Epidural steroid injection (Other)
  Interventions: Other: Epidural steroid injection

INTERVENTIONS:
Other: Epidural steroid injection plus physical therapy — Patients in the ESI+PT Group will be treated additionally with a physical therapy program emphasizing lumbar flexion exercises, aerobic and strength/ conditioning exercises, and manual physical therapy as well as receiving up to 3 epidural steroid injection(s) and educational support using The Back Book.
  Arms: Epidural steroid injection and physical therapy
Other: Epidural steroid injection — Patients in the ESI Group will be treated with up to 3 epidural steroid injections, educational support, and general care by the treating physician.
  Arms: Epidural steroid injection

SUMMARY:
Lumbar spinal stenosis (LSS) is a prevalent and disabling condition in the rapidly growing aging population. People with LSS often have a substantial physical and psychosocial burden as well as significant healthcare costs affecting both the individual and society. It has been reported that patients with LSS over the age of 65 are more likely to undergo spinal surgery than any other condition with an estimated total annual inpatient expense of one billion. Individuals undergoing surgical treatment for LSS tend to be older, therefore operative morbidity and mortality are a particular concern. Functional benefit derived from conservative treatment may increase the health and quality of life for individuals suffering from LSS and avoid or delay the need for surgery in some subjects. As the population continues to age, identifying effective non-surgical treatment options for older patients with LSS is an important research priority. Ultimately, the information gained from this study will help fill a significant void in medical literature regarding non-surgical options for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Lumbar spinal stenosis unidentified by MRI or CT scan and interpreted by a radiologist independent of the study. The criteria of Boden et al will be used to define LSS on MRI: non-discogenic loss of signal in the epidural fat with compression of neural tissues.
2. Chief complaint of pain in the low back, buttock, and/or lower extremity. The patient must have LE symptoms consistent with neurogenic claudiation.
3. Patient-reported inability to walk greater than ¼ mile due to lower extremity pain and/or cramping.
4. Rates sitting as a better position with respect to symptom severity compared to standing or walking.
5. Consent of the patient to undergo education, epidural steroid injection(s), and attend specified physical therapy sessions.
6. Individuals with no language barrier, that are cooperative, have transportation to the Spine Center, and who sign an informed consent form.
7. Age greater than or equal to 50 years.

Exclusion Criteria:

1. Patients with organic brain syndrome or dementia.
2. Severe vascular, pulmonary or coronary artery disease which limits ambulation.
3. Recent myocardial infarction (within last 6 months).
4. Spondylolisthesis requiring surgical fusion (i.e., greater than 5mm of slippage).
5. Previous spinal surgery that included fusion of two or more vertebrae.
6. Severe osteoporosis as defined by multiple compression fractures or a fracture at the same level as the stenosis.
7. Metastatic cancer.
8. Excessive alcohol consumption or evidence of non-prescribed or illegal drug use.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest will be change in disability as measured by the Modified Oswestry Disability Index (OSW). | 10 weeks, 6 months, 12 months

SECONDARY OUTCOMES:
Change in patient-reported pain | 10 weeks, 6 months, 12 months
Change in Functional Limitations | 10 weeks, 6 months, 12 months
Change in psychosocial evaluation | 10 weeks, 6 months, 12 months
Change in patient satisfaction | 10 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Colorado University, Denver, Colorado
  - Illinois Neurological Institute at OSF, Peoria, Illinois
  - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Hawkins Foundation, Greenville, South Carolina

REFERENCES:
- [Derived] Hammerich A, Whitman J, Mintken P, Denninger T, Akuthota V, Sawyer EE, Hofmann M, Childs JD, Cleland J. Effectiveness of Physical Therapy Combined With Epidural Steroid Injection for Individuals With Lumbar Spinal Stenosis: A Randomized Parallel-Group Trial. Arch Phys Med Rehabil. 2019 May;100(5):797-810. doi: 10.1016/j.apmr.2018.12.035. Epub 2019 Jan 29. PMID 30703349